CLINICAL TRIAL: NCT02207478
Title: Diagnostic Value of Electromagnetic Navigation Bronchoscopy With a Guide Sheath for Peripheral Pulmonary Lesions : a Randomized Controlled Trial
Brief Title: ENB-GS-TBLB for the Diagnosis of PPLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Endoscope Center, Shanghai Chest Hospita, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHCHE201401
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer
Keywords: Electromagnetic navigation bronchoscopy with a guide sheath; Transbronchial lung biopsy; Peripheral lung lesions; Solitary pulmonary nodule
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ENB-GS-TBLB-X-ray Group (Experimental): The guide sheath(GS) is introduced into the lesion via Electromagnetic Navigation System. The locatable guide(LG) and GS are confirmed to reach the lesion by radiograph fluoroscopy, pathologic specimens are obtained with fluoroscopic guidance.
  Interventions: Procedure: ENB; Procedure: GS-TBLB-X-ray
- GS-TBLB-X-ray group (Active Comparator): The GS is introduced into the lesion via the working channel of a bronchoscope with radiographic fluoroscopy. Once the location of the lesion is identified by fluoroscopy, pathologic specimens are obtained under fluoroscopic guidance.
  Interventions: Procedure: GS-TBLB-X-ray

INTERVENTIONS:
Procedure: ENB — ENB is performed using an electromagnetic navigation system (LK-DW-NK-Z; Suzhou Lungcare Medical Technology Inc., China) with an internal locatable guide (LG; Lungcare) with diameter of 1.45 mm. Bronchoscopes with a working channel diameter of 2.0 mm are used (BF-260 and BF-P260F; Olympus, Japan). The LG is inserted into the GS(K-201; Olympus) beforehand, and the GS-covered LG is introduced via the working channel of the bronchoscope and navigated to the PPL finally. The LG and GS are confirmed to reach the lesion by radiograph fluoroscopy.
  Arms: ENB-GS-TBLB-X-ray Group
Procedure: GS-TBLB-X-ray — A GS is introduced in the working channel of the bronchoscope alone. The GS is confirmed to reach the lesion by radiograph fluoroscopy, pathologic specimens are obtained under fluoroscopic guidance.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of electromagnetic navigation bronchoscopy with a Guide Sheath(ENB-GS) for the diagnosis of peripheral pulmonary lesions (PPLs) .

DETAILED DESCRIPTION:
The investigators evaluated the efficacy and safety of transbronchial lung biopsy (TBLB) and bronchial brushing using electromagnetic navigation bronchoscopy (ENB) with a guide sheath (GS) for the diagnosis of peripheral pulmonary lesions (PPLs) with radiographic fluoroscopy.The study is designed as a two-center prospective randomized controlled trial. The participating centers are Department of pulmonary medicine and endoscope department, Shanghai chest Hospital affiliated to Shanghai JiaoTong University, China. Department of pulmonary medicine, Shanghai ZhongShan Hospitial affiliated to Shanghai FuDan University, China.Patients are divided into two groups, ENB-GS-TBLB-X-ray group and GS-TBLB-X-ray group.Each subject will be randomized to each group.The study is expected to enroll 60 patients at 2 centers (Shanghai Chest Hospital: 40, Shanghai Zhongshan Hospital: 20).

ELIGIBILITY:
Inclusion Criteria:

1. clinical and imaging characteristics suggestive of maligancy
2. CT scan appearance of the PPLs showed the longest diameter was more than 1 cm and solid lesions.

Exclusion Criteria:

1. The lesion is close to the pleural membrane
2. Refusal of participation
3. Severe cardiopulmonary dysfunction and other indications that can't receive bronchoscopy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

REFERENCES:
- [Background] Gex G, Pralong JA, Combescure C, Seijo L, Rochat T, Soccal PM. Diagnostic yield and safety of electromagnetic navigation bronchoscopy for lung nodules: a systematic review and meta-analysis. Respiration. 2014;87(2):165-76. doi: 10.1159/000355710. Epub 2014 Jan 3. PMID 24401166
- [Background] Baaklini WA, Reinoso MA, Gorin AB, Sharafkaneh A, Manian P. Diagnostic yield of fiberoptic bronchoscopy in evaluating solitary pulmonary nodules. Chest. 2000 Apr;117(4):1049-54. doi: 10.1378/chest.117.4.1049. PMID 10767238
- [Background] Wang Memoli JS, Nietert PJ, Silvestri GA. Meta-analysis of guided bronchoscopy for the evaluation of the pulmonary nodule. Chest. 2012 Aug;142(2):385-393. doi: 10.1378/chest.11-1764. PMID 21980059

RESULTS

PARTICIPANT FLOW:
Groups:
- ENB-GS-TBLB-X-ray Group: The guide sheath(GS) is introduced into the lesion via Electromagnetic Navigation System.
  ENB: ENB is performed using an electromagnetic navigation system (LK-DW-NK-Z; Suzhou Lungcare Medical Technology Inc., China) with an internal locatable guide (LG; Lungcare) with diameter of 1.45 mm. Bronchoscopes with a working channel diameter of 2.0 mm are used (BF-260 and BF-P260F; Olympus, Japan). The LG is inserted into the GS(K-201; Olympus) beforehand, and the GS-covered LG is introduced via the working channel of the bronchoscope and navigated to the PPL finally. The LG and GS are confirmed to reach the lesion by radiograph fluoroscopy.
  GS-TBLB-X-ray: A GS is introduced in the working channel of the bronchoscope alone. The GS is confirmed to reach the lesion by radiograph fluoroscopy, pathologic specimens are obtained under fluoroscopic guidance.
Period: Overall Study
Arm/Group | ENB-GS-TBLB-X-ray Group | GS-TBLB-X-ray Group
Started | 40 | 46
Completed | 40 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ENB-GS-TBLB-X-ray Group | GS-TBLB-X-ray Group | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.28 (7.61) | 59.32 (9.57) | 60.28 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 20 | 27 | 47
lesion size(long axis) [Mean (Standard Deviation); unit: mm] | 29.7 (11) | 33.07 (13.8) | 31.39 (12.51)
lesion size(short axis) [Mean (Standard Deviation); unit: mm] | 21.64 (10.42) | 22.28 (10.66) | 21.96 (10.47)
lesion location [Number; unit: participants]
  Upper Lobes | 26 | 29 | 55
  Middle Lobes | 3 | 1 | 4
  Lower lobes | 10 | 11 | 21
distance from the lesion to the pleural [Mean (Standard Deviation); unit: mm] — distance of the nodule to the pleural surface
  mm | 15.53 (14.79) | 20.99 (16.08) | 18.19 (15.57)
bronchus sign [Number; unit: participants] — The bronchus sign on CT represents the presence of a bronchus leading directly to a peripheral pulmonary lesion.
  participants
    Yes | 32 | 38 | 70
    No | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: The Difference of Diagnostic Value of ENB-GS-TBLB as Compared to GS-TBLB
Description: The diagnostic yield in the ENB-GS-TBLB and GS-TBLB group was 87.2% and 61% individually.
Time Frame: Up to half year
Measure: Number; unit: participants
Arm/Group | ENB-GS-TBLB-X-ray Group | GS-TBLB-X-ray Group
Number analyzed (Participants) | 39 | 41
participants
  Diagnosed by TBLB | 34 | 25
  Not Diagnosed by TBLB | 5 | 16
Statistical Analysis 1: Comparison: ENB-GS-TBLB-X-ray Group vs GS-TBLB-X-ray Group; Test type: Superiority or Other; p = 0.019, Cochran-Mantel-Haenszel

2. Secondary Outcome: The Duration Time Difference of ENB-GS-TBLB With Fluoroscopy as Compared to GS-TBLB With Fluoroscopy Alone
Description: Including total procedure time，total X-ray time, duration time for finding lesions and X-ray time for finding lesions.
Time Frame: Up to half year
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | ENB-GS-TBLB-X-ray Group | GS-TBLB-X-ray Group
Number analyzed (Participants) | 39 | 41
seconds
  Total procedure time | 1053.6 (408.6) | 1056.6 (387)
  Total X-ray time | 156.56 (94.03) | 142.27 (111.84)
  Duration time for finding lesion | 126.74 (128.80) | 224.98 (119.08)
  X-ray time for finding lesion | 7.21 (7.79) | 38.88 (39.37)
Statistical Analysis 1: Comparison: ENB-GS-TBLB-X-ray Group vs GS-TBLB-X-ray Group; Total procedure time; Test type: Superiority or Other; p = 0.843, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ENB-GS-TBLB-X-ray Group vs GS-TBLB-X-ray Group; Total X-ray time; Test type: Superiority or Other; p = 0.233, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ENB-GS-TBLB-X-ray Group vs GS-TBLB-X-ray Group; Duration time for finding lesions; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: ENB-GS-TBLB-X-ray Group vs GS-TBLB-X-ray Group; X-ray time for finding lesions; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | ENB-GS-TBLB-X-ray Group | GS-TBLB-X-ray Group
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/41
Other Adverse Events (participants affected / at risk) | 0/39 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No